CLINICAL TRIAL: NCT07184099
Title: Effect of Phloroglucinol on Shortening the Duration of Active Phase of Labor
Brief Title: Phloroglucinol Effectiveness on Shortening the Duration of Active Phase of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Tahira-Attock
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Labor
MeSH Terms: interventions — Phloroglucinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phloroglucinol group (Experimental): Phloroglucinol was administered as intravenous stat infusion with Ringer Lactate infusion.
  Interventions: Drug: Phloroglucinol
- Placebo group (No Intervention): The patients were given only Ringer Lactate infusion.

INTERVENTIONS:
Drug: Phloroglucinol — Phloroglucinol was administered as intravenous stat infusion with Ringer Lactate infusion.
  Arms: Phloroglucinol group

SUMMARY:
This study was planned to fill the gaps regarding the effectiveness of phloroglucinol on the duration of active phase of labor.

DETAILED DESCRIPTION:
In today's era, the focus has shifted from a "wait and watch" policy to "active intervention sooner than later" to enhance better labor outcomes. Using an ideal antispasmodic drug would help achieve a rapid and prolonged effect on cervical dilation, with no adverse impact on uterine contractions or causing uterine inertia. If the current study finds phloroglucinol effective in shortening the duration of the active phase of labor, it would help achieve better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged between 18-35 years
* Period of gestation above 37 weeks.

Exclusion Criteria:

* Women with cephalopelvic disproportion
* Double scare uterus
* Fetal distress
* Life threatening bleeding
* Eclampsia
* History of heart disease
* Known allergy to phloroglucinol

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Duration of labor | 4 hours
  The duration of labor was measured from the time of diagnosis of labor until full dilatation of cervix.

CONTACTS AND LOCATIONS:
Overall Officials: Tahira Riaz, FCPS, Principal Investigator — Combined military hospital Attock
Locations (1):
- Combined Military Hospital, Attock, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.